CLINICAL TRIAL: NCT05744115
Title: Utility of Ga-68-PSMA-11 in Management of Prostate Cancer
Brief Title: Ga-68-PSMA-11 in Men With Prostate Cancer
Acronym: Ga68-PSMA-11
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The investigational product was approved by the FDA (12/20/2021) and is now commercially available
Sponsor: Timothy Hoffman (U.S. Federal Agency)
Collaborators: Harry S. Truman Memorial Veterans' Hospital (U.S. Federal Agency); University of Missouri-Columbia (Other); Telix Pharmaceuticals, Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Timothy Hoffman, Research Career Scientist, Harry S. Truman Memorial Veterans' Hospital
Organization: Harry S. Truman Memorial Veterans' Hospital (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2031231
Record Dates: First submitted 2023-02-01; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
Keywords: PSMA; Biochemically Recurrent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Intervention Model Description: All eligible and consenting participants (male veterans) will receive a single administration of 3-7mCi Ga-68-PSMA-11 per enrollment in addition to conventional imaging (MRI, CT, and/or molecular imaging bone scan).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ga-68-PSMA-11 PET/CT (Experimental): Administration of Ga-68-PSMA-11 and acquisition of PET/CT
  Interventions: Drug: Ga-68-PSMA-11

INTERVENTIONS:
Drug: Ga-68-PSMA-11 — Ga-68-PSMA-11 is produced via a lyophilized Sterile Cold kit. Ga-68 is eluted from a Ge-68/Ga-68 generator into a vial containing the premixed peptide and buffer. PSMA-11 radiolabeled with Ga-68 is administered to patients following verification of standard quality controls including activity measurement, pH, radiochemical purity, and visual inspection

SUMMARY:
The purpose of this study is to provide access to Ga-68-PSMA-11 PET for evaluation of male veterans with newly diagnosed or biochemically recurrent prostate cancer. All patients will receive conventional imaging (MRI, CT, and/or a molecular imaging bone scan) as well as Ga-68-PSMA-11 PET in order to evaluate the utility of diagnostic testing in patients with positive PSA status, a comparison of results from conventional imaging and PSMA PET imagining will be performed.

DETAILED DESCRIPTION:
Participants (male veterans) with initial diagnosis of prostate cancer or biochemically recurrent disease that consent to participate in the study will receive both conventional imaging (MRI, CT, and/or molecular imaging bone scan) as well as Ga-68-PSMA-11 PET/CT. Following baseline assessment (Visit #1), Ga-68-PSMA-11 (3-7 mCi) will be administered as a single intravenous administration with PET/CT performed approximately 60 minutes after injection (Visit #2A). At approximately 120 minutes after injection of Ga-68-PSMA-11, the final evaluation for safety and tolerability will occur (Visit #2B)

ELIGIBILITY:
Inclusion Criteria:

* Able to tolerate PET/CT imaging and one or more of the following:
* Patients with newly diagnosed prostate cancer with primary staging classified at high/intermediate risk per NCCN guidelines OR
* Biochemical Recurrence: Patients with rising PSA after definitive therapy with prostatectomy or radiation therapy or other local therapies

Exclusion Criteria:

* Claustrophobia or any other condition that would preclude PET/CT imaging.
* Any constellation of medical conditions that indicate expectancy of less than one year

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male Veterans over the age of 18 years with previously diagnosed prostate cancer
Enrollment: 38 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Concurrence with Conventional Imaging | Up to 28 days
  Localized vs extra-pelvic recurrence will be determined for each patient based on Ga-68-PSMA-11 PET/CT and standard-of-care radiological imaging

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Hoffman, PhD, Principal Investigator — Truman VA Hospital; Columbia, MO
Locations (1):
- Truman VA Hospital, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be prepared to share with other VA investigators upon request